CLINICAL TRIAL: NCT01746953
Title: The Effect of Red Blood Cells Transfusion in Trauma Patients: A Risk Stratified Analysis
Brief Title: The Effect of Red Blood Cells Transfusion in Trauma Patients
Status: Completed | Type: Observational
Sponsor: Progress (Network)
Responsible Party: Sponsor
Other Study IDs: Progress-06; G0902393/99558 (Other Grant/Funding Number: MRC)
Record Dates: First submitted 2012-12-07; First posted 2012-12-11 (Estimated); Last update posted 2012-12-11 (Estimated); Status verified 2012-12

CONDITIONS: Trauma
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
We will evaluate the effect of red blood cell (RBC) transfusion on fatal and non fatal events according to baseline risk of death in an international cohort of trauma patients (CRASH-2 trial). The following outcomes will be considered: death from all causes, death due to bleeding, death due to multiorgan failure, death due to vascular occlusive events and non vascular occlusive events. Non fatal outcomes include: myocardial infarction, stroke, deep vein thrombosis and pulmonary embolism.

DETAILED DESCRIPTION:
Aims: Primary objective: Evaluate the effect of RBC transfusion on all cause mortality according to baseline risk of death due to bleeding. Secondary objectives: Evaluate the effect of RBC transfusion on specific causes of death. Evaluate the effect of RBC transfusion on non fatal vascular occlusive events.

Sample: Patients from the Clinical Randomisation of an Antiﬁbrinolytic in Signiﬁcant Haemorrhage (CRASH-2) trial. The trial included 20,127 trauma patients with, or at risk of, significant bleeding, within 8 hours of injury, and was undertaken in 274 hospitals in 40 countries.

Outcomes: Death from all causes, death due to bleeding, death due to multiorgan failure, death due to vascular occlusive events and non vascular occlusive events. Vascular occlusive events include: myocardial infarction, stroke, deep vein thrombosis and pulmonary embolism. All events were measured at 28 days or hospital discharge Interventions and comparisons: We will compare the effect of red cells transfusion versus no red cells transfusion. We will also evaluate the effect of the number of units of red cells transfusion.

Methods: We will stratify patients according to baseline risk of death from all causes into four strata (<6%, 6%-20%, 21%-50% and >50%). We will then evaluate the effect of RBC transfusion according to baseline risk on fatal and non fatal outcomes. Formal statistical test to detect heterogeneity will be conducted analyzing baseline risk as a continuous variable.

ELIGIBILITY:
Inclusion Criteria:

* Patients eligible for inclusion in the trial were "adult trauma patients with ongoing significant haemorrhage, within 8 hours of injury."

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from the Clinical Randomisation of an Antiﬁbrinolytic in Signiﬁcant Haemorrhage (CRASH-2) trial. The trial included 20,127 trauma patients with, or at risk of, significant bleeding, within 8 hours of injury, and was undertaken in 274 hospitals in 40 countries.
Sampling Method: Non-Probability Sample
Enrollment: 20211 (Actual)
Dates: Start 2005-05; Primary Completion 2010-02 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
mortality | 30 days

SECONDARY OUTCOMES:
fatal and non fatal vascular occlusive events | 30 days

REFERENCES:
- [Derived] Perel P, Clayton T, Altman DG, Croft P, Douglas I, Hemingway H, Hingorani A, Morley KI, Riley R, Timmis A, Van der Windt D, Roberts I; PROGRESS Partnership. Red blood cell transfusion and mortality in trauma patients: risk-stratified analysis of an observational study. PLoS Med. 2014 Jun 17;11(6):e1001664. doi: 10.1371/journal.pmed.1001664. eCollection 2014 Jun. PMID 24937305